CLINICAL TRIAL: NCT06176196
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel-design Study of the Efficacy and Safety of VX-548 in Subjects With Painful Lumbosacral Radiculopathy
Brief Title: Evaluation of Efficacy and Safety of VX-548 for Painful Lumbosacral Radiculopathy (PLSR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX23-548-109
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Painful Lumbosacral Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VX-548 (Experimental): Participants will receive VX-548 up to 12 weeks.
  Interventions: Drug: VX-548
- Placebo (Placebo Comparator): Participants will receive placebo matched to VX-548 up to 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-548 — Tablets for oral administration.
  Other Names: Suzetrigine
  Arms: VX-548
Drug: Placebo — Tablets for oral administration.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of VX-548 in treating participants with PLSR.

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight greater than or equal to (>=)45 kilogram (kg)
* Body mass index (BMI) less than or equal to (<=) 40 kg/ meter square (m^2)
* Diagnosis of PLSR for greater than (>)3 months as per criteria pre-specified in the protocol
* Weekly average of daily NPRS score >=4 and <10 with limited variation in the 7-day Run-in Period

Key Exclusion Criteria:

* More than 3 missing daily NPRS scores during the 7-day Run-in Period
* Moderate or severe painful neuropathy other than PLSR as pre-specified in the protocol
* History of prior lumbar spine surgery (e.g., discectomies, laminectomies, foraminotomies, or fusion)

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in the Weekly Average of Daily leg Pain Intensity on a Numeric Pain Rating Scale (NPRS) | Baseline, Week 12

SECONDARY OUTCOMES:
Change From Baseline in the Weekly Average of the Daily Sleep Interference Scale (DSIS) | Baseline, Week 12
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Week 14

CONTACTS AND LOCATIONS:
Locations (54):
- United States (54):
  - Hope Research Institute, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Trovare Clinical Research, Bakersfield, California
  - Velocity Clinical Research - Banning, Banning, California
  - Velocity Clinical Research - San Diego, La Mesa, California
  - Probe Clinical Research, Riverside, California
  - Pain Management and Injury Relief, Thousand Oaks, California
  - Visionary Investigators Network, Aventura, Florida
  - Nature Coast Clinical Research - Crystal River, Crystal River, Florida
  - JY Research Institute, Cutler Bay, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Convenient Medical Research, Hialeah, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - L&C Professional Medical Research Institute, Miami, Florida
  - Medical Research of Westchester, Miami, Florida
  - ARSN-Brain and Spine Institute, Port Orange, Florida
  - Accel Research Site - St. Petersburg/Largo, Seminole, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - ClinCept Clinical Research, Columbus, Georgia
  - Accel Research Sites - Neurostudies, Decatur, Georgia
  - Velocity Clinical Research - Savannah Neurology Specialists, Savannah, Georgia
  - Velocity Clinical Research - Savannah, Savannah, Georgia
  - Center for Pain Management and Rehab, Stockbridge, Georgia
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Healthcare Research Network II, LLC, Flossmoor, Illinois
  - Essential Concepts Research Solutions, Palos Hills, Illinois
  - AMR Wichita East, KS, Wichita, Kansas
  - Velocity Clinical Research - Rockville, Rockville, Maryland
  - Brigham and Women's Hospital (BWH), Boston, Massachusetts
  - MedVadis Research Coorporation, Waltham, Massachusetts
  - St. Louis Pain Consultants, Chesterfield, Missouri
  - Healthcare Research Network, Hazelwood, Missouri
  - Be Well Clinical Studies, LLC, Lincoln, Nebraska
  - Synexus Clinical Research - Henderson, Henderson, Nevada
  - AMR Las Vegas (Clinical Research Consortium), Las Vegas, Nevada
  - Albany Medical Center, Albany, New York
  - AES New York, New York, New York
  - Velocity Clinical Research - Cincinnati, Cincinnati, Ohio
  - META Medical Research Institute, Dayton, Ohio
  - NexGen Research, Lima, Ohio
  - Clinical Investigations LLC., Edmond, Oklahoma
  - AMR Norman, Norman, Oklahoma
  - Pacific Sports and Spine, Eugene, Oregon
  - Velocity Clinical Research - Grants Pass, Grants Pass, Oregon
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - Clinical Trials of South Carolina - Charleston, Charleston, South Carolina
  - AES Dallas Forth Worth, Dallas, Texas
  - Expert Pain, Houston, Texas
  - Lubbock Spine Institute, Lubbock, Texas
  - Be Well Clinical Studies - Austin, Round Rock, Texas
  - JBR Clinical Research, Salt Lake City, Utah
  - Velocity Clinical Research - Hampton, Hampton, Virginia
  - AMR Norfolk, Norfolk, Virginia
  - Velocity Clinical Research - Portsmouth, Portsmouth, Virginia

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Siddiqui A, Xu JL, Abramowicz AE. Suzetrigine for the Treatment of Acute Pain: Comment. Anesthesiology. 2026 Feb 1;144(2):495-496. doi: 10.1097/ALN.0000000000005822. Epub 2025 Dec 11. No abstract available. PMID 41384808